CLINICAL TRIAL: NCT02902068
Title: Maternal Hemodynamic Monitoring in Women Undergoing Cesarean Section by Use of NICaS Cardiac Impedance
Brief Title: Hemodynamic Monitoring in Women Throughout Cesarean Sections
Status: Completed | Type: Observational
Sponsor: Rabin Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 0512-15-RMC
Record Dates: First submitted 2016-06-01; First posted 2016-09-15 (Estimated); Last update posted 2019-03-29 (Actual); Status verified 2016-05

CONDITIONS: Hemodynamics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Parturients undergoing cesarean section: Healthy parturients, hypertensive parturients and parturients suffering from preeclampsia above 18 undergoing cesarean section deliveries .
  Interventions: Device: NICaS Bio Impedance

INTERVENTIONS:
Device: NICaS Bio Impedance — Hemodynamic monitoring will be carried out using non invasive NICaS cardiac impedance by the use of two electrodes stickers which are pasted on the wrists for about 6 minutes.
  Monitoring will be done with women lying down or sitting up half an hour preoperatively (in the woman's surgery waiting room) intraoperatively, and postoperatively in the PACU.
  Preoperative data will be compared to intraoperative and postoperative data, and will be analyzed in order to evaluate the dynamic cardiac output changes in women undergoing cesarean sections.

SUMMARY:
In this study we would like to monitor cardiac output by the use of NICAS bioimpedance in women undergoing cesarean section delivery.

This study is a purely observational study, it will not have any clinical intervention nor will it interfere with standard cesarean delivery protocols in any way. This study's primary objective is to evaluate how spinal and general anesthesia influences cardiac output during cesarean section deliveries. Secondary endpoints is whether the hemodynamic changes as measured in cardiac output correlate with women's pain, measured by a visual analogue scale(VAS) from o-10. (0=representing no pain at all, 10= worse pain imaginable)

DETAILED DESCRIPTION:
This is a prospective, single center study which will be conducted at the Rabin Medical Center (Beilinson Campus), Petach Tikva, Israel, a tertiary university hospital. The Institutional Review Board has approved this study.

Two hundred women undergoing cesarean sections will be enrolled after filling out an informed consent form. Women will be recruited half an hour preoperatively in the women's surgery waiting room when they aren't experiencing any pain, and aren't under any sedatives.

Following obtaining an informed consent maternal cardiac output will be monitored.

The monitoring will be carried out using non invasive NICaS cardiac impedance by the use of two electrodes stickers which are pasted on the wrists for about 6 minutes.

Monitoring will be done with women lying down or sitting up half an hour preoperatively (in the woman's surgery waiting room) intraoperatively, and postoperatively in the post anesthesia care unit (PACU).

Preoperative data will be compared to intraoperative and postoperative data, and will be analyzed in order to evaluate the dynamic cardiac output changes in women undergoing cesarean sections.

Recorded data will include:

* Demographic and obstetric - age, weight, height, current hemoglobin, co-morbidities, regular medication and other obstetric data.
* Cardiovascular risk factors - a family history of cardiovascular disease, smoking, BMI
* Obstetric history - obstetric background (history of gestational diabetes, preeclampsia, intrauterine growth restriction (IUGR), stillbirths or placental abruption).
* Threshold of pain according to VAS It should be emphasized that the conduct of the study will not interfere in with cesarean delivery protocol in any way.

ELIGIBILITY:
Inclusion Criteria:

- All women undergoing cesarean section in Beilinson Hospital following obtaining written informed consents forums with the ability to comply to the study requirements will be included in our study.

Exclusion Criteria:

- Women under age 18 , and women who don't understand the inform consent form will be excluded from participating.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy and hypertensive women above 18 undergoing cesarean section deliveries.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2016-05; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Hemodynamic changes in cesarean section as measured by NICaS parameters. | A year
  This study's primary objective is to evaluate how anesthesia influences cardiac output during cesarean section deliveries

SECONDARY OUTCOMES:
Hemodynamic changes measured by NICaS parameters and their correlation with pain in women undergoing cesarean sections as measured by VAS. | A year

CONTACTS AND LOCATIONS:
Locations (1):
- Beilinson hospital, Petach Tikvah, Israel

IPD SHARING:
Plan to Share IPD: Undecided
In this study the investigators would like to monitor cardiac output by the use of NICaS bioimpedance in women undergoing cesarean section delivery.
  This study is a purely observational study, it will not have any clinical intervention nor will it interfere with standard cesarean delivery protocols in any way.

REFERENCES:
- [Background] Dennis AT, Dyer RA. Cardiac output monitoring in obstetric anaesthesia. Int J Obstet Anesth. 2014 Feb;23(1):1-3. doi: 10.1016/j.ijoa.2013.11.001. Epub 2013 Nov 13. No abstract available. PMID 24300387
- [Background] Bliacheriene F, Carmona MJ, Barretti Cde F, Haddad CM, Mouchalwat ES, Bortolotto MR, Francisco RP, Zugaib M. Use of a minimally invasive uncalibrated cardiac output monitor in patients undergoing cesarean section under spinal anesthesia: report of four cases. Rev Bras Anestesiol. 2011 Sep-Oct;61(5):610-8, 334-8. doi: 10.1016/S0034-7094(11)70072-1. English, Portuguese, Spanish. PMID 21920211
- [Background] Dyer RA, James MF. Maternal hemodynamic monitoring in obstetric anesthesia. Anesthesiology. 2008 Nov;109(5):765-7. doi: 10.1097/ALN.0b013e31818a3825. No abstract available. PMID 18946283
- [Background] Langesaeter E. Is it more informative to focus on cardiac output than blood pressure during spinal anesthesia for cesarean delivery in women with severe preeclampsia? Anesthesiology. 2008 May;108(5):771-2. doi: 10.1097/ALN.0b013e31816bbe04. No abstract available. PMID 18431110
- [Background] Langesaeter E, Gibbs M, Dyer RA. The role of cardiac output monitoring in obstetric anesthesia. Curr Opin Anaesthesiol. 2015 Jun;28(3):247-53. doi: 10.1097/ACO.0000000000000190. PMID 25915203
- [Background] Dyer RA, Reed AR, van Dyk D, Arcache MJ, Hodges O, Lombard CJ, Greenwood J, James MF. Hemodynamic effects of ephedrine, phenylephrine, and the coadministration of phenylephrine with oxytocin during spinal anesthesia for elective cesarean delivery. Anesthesiology. 2009 Oct;111(4):753-65. doi: 10.1097/ALN.0b013e3181b437e0. PMID 19741494
- [Background] Langesaeter E, Rosseland LA, Stubhaug A. Continuous invasive blood pressure and cardiac output monitoring during cesarean delivery: a randomized, double-blind comparison of low-dose versus high-dose spinal anesthesia with intravenous phenylephrine or placebo infusion. Anesthesiology. 2008 Nov;109(5):856-63. doi: 10.1097/ALN.0b013e31818a401f. PMID 18946298
- [Background] Habib AS. A review of the impact of phenylephrine administration on maternal hemodynamics and maternal and neonatal outcomes in women undergoing cesarean delivery under spinal anesthesia. Anesth Analg. 2012 Feb;114(2):377-90. doi: 10.1213/ANE.0b013e3182373a3e. Epub 2011 Nov 21. PMID 22104076
- [Background] Langesaeter E, Dyer RA. Maternal haemodynamic changes during spinal anaesthesia for caesarean section. Curr Opin Anaesthesiol. 2011 Jun;24(3):242-8. doi: 10.1097/ACO.0b013e32834588c5. PMID 21415724
- [Background] Tihtonen K, Koobi T, Yli-Hankala A, Huhtala H, Uotila J. Maternal haemodynamics in pre-eclampsia compared with normal pregnancy during caesarean delivery. BJOG. 2006 Jun;113(6):657-63. doi: 10.1111/j.1471-0528.2006.00931.x. PMID 16709208
- [Background] Melchiorre K, Sutherland GR, Baltabaeva A, Liberati M, Thilaganathan B. Maternal cardiac dysfunction and remodeling in women with preeclampsia at term. Hypertension. 2011 Jan;57(1):85-93. doi: 10.1161/HYPERTENSIONAHA.110.162321. Epub 2010 Nov 22. PMID 21098311
- [Background] McDonald SD, Malinowski A, Zhou Q, Yusuf S, Devereaux PJ. Cardiovascular sequelae of preeclampsia/eclampsia: a systematic review and meta-analyses. Am Heart J. 2008 Nov;156(5):918-30. doi: 10.1016/j.ahj.2008.06.042. Epub 2008 Oct 2. PMID 19061708
- [Background] Dyer RA, Piercy JL, Reed AR, Lombard CJ, Schoeman LK, James MF. Hemodynamic changes associated with spinal anesthesia for cesarean delivery in severe preeclampsia. Anesthesiology. 2008 May;108(5):802-11. doi: 10.1097/01.anes.0000311153.84687.c7. PMID 18431115
- [Background] Critchley LA, Lee A, Ho AM. A critical review of the ability of continuous cardiac output monitors to measure trends in cardiac output. Anesth Analg. 2010 Nov;111(5):1180-92. doi: 10.1213/ANE.0b013e3181f08a5b. Epub 2010 Aug 24. PMID 20736431
- [Background] Critchley LA, Critchley JA. A meta-analysis of studies using bias and precision statistics to compare cardiac output measurement techniques. J Clin Monit Comput. 1999 Feb;15(2):85-91. doi: 10.1023/a:1009982611386. PMID 12578081
- [Background] Chaffin DG, Webb DG. Outcomes of pregnancies at risk for hypertensive complications managed using impedance cardiography. Am J Perinatol. 2009 Nov;26(10):717-21. doi: 10.1055/s-0029-1223283. Epub 2009 May 18. PMID 19452431